CLINICAL TRIAL: NCT03879577
Title: Assessing REsponse to Neoadjuvant Taxotere and Trastuzumab in Nigerian Women With HER2-positive Breast Cancer (ARETTA)
Brief Title: Assessing the Response Rate of Neo-adjuvant Taxotere and Trastuzumab in Nigerian Women With Breast Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB18-1178
Record Dates: First submitted 2019-02-12; First posted 2019-03-19 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-08

CONDITIONS: Breast Cancer; Breast Cancer Female; HER2-positive Breast Cancer; Breast Cancer Stage II; Breast Cancer Stage III
Keywords: breast cancer; breast cancer stage II; Breast Cancer Stage III; Docetaxel; Herceptin; neoadjuvant treatment; nigeria
MeSH Terms: conditions — Breast Neoplasms | interventions — Docetaxel; Trastuzumab; Tamoxifen; Letrozole; Gonadotropin-Releasing Hormone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Neoadjuvant taxotere and trastuzumab (Experimental): Investigators will give patients docetaxel/taxotere through drip every 3 weeks for four doses for 12 weeks before a repeat breast ultrasound. After breast ultrasound, if the investigator feels the injection is good, surgery will be done.
  Herceptin/trastuzumab will be given to patients under the skin of the thigh every 3 weeks for 18 times if they are HER2-positive
  Patients with a poor response to docetaxal/herceptin will receive Fluorouracil, Epirubicin Hydrochloride, Cyclophonsphamide (FEC) injection by drip every 3 weeks.
  Hormone-receptor positive patients will receive hormonal therapy with tamoxifen or letrozole after surgery, radiotherapy and LHRH agonist according to the expression of hormone receptors and according to the state of primary menopause at the onset of the study.
  Interventions: Drug: Docetaxel; Drug: Herceptin; Drug: FEC; Drug: Tamoxifen; Drug: Letrozole; Drug: LHRH agonist

INTERVENTIONS:
Drug: Docetaxel — Administered to all patients for a minimum of 4 cycles for 12 weeks.
Drug: Herceptin — Administered for 18 cycles every three weeks (52 weeks) for each patient starting at the first day of treatment with docetaxel.
  Other Names: Trastuzumab
Drug: FEC — Only administered to patients who received docetaxel and herceptin and were assessed as having poor response (defined as stable disease or progressive disease or partial response inoperable).
Drug: Tamoxifen — Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
Drug: Letrozole — Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
Drug: LHRH agonist — Administered to all premenopausal patients.

SUMMARY:
This is a one stage phase II study with a single arm design. It will be conducted in HER-2 positive breast cancer patients in Nigeria who are chemotherapy/hormonal treatment naive.

ELIGIBILITY:
Inclusion Criteria:

1. Women ages of 18 to 70 years old
2. Biopsy-accessible breast tumor of significant size for core needle biopsy/ultrasound measurable (≥ 2cm)
3. Patients with histologically confirmed carcinoma of the female breast with 3+ positive HER2 status by IHC
4. Clinical stages IIA -IIIC (AJCC 2009)
5. Chemotherapy-naïve patients (for this malignancy)
6. Performance status: ECOG performance status 0-1 (Appendix A)
7. Non-pregnant and not nursing. Women of childbearing potential must take the pregnancy test and must commit to receive LHRH agonist Zoladex (goserelin) for two years starting from the commencement of the study medications
8. Required Initial Laboratory Data. Adequate hematologic, renal and hepatic function, as defined by each of the following:

1. Granulocyte ≥ 1,500/μL 2. Platelet count ≥ 100,000/μL 3. Absolute neutrophil count (ANC) ≥ l500/μL 4. Hemoglobin ≥ 10g/dL 5. Bilirubin ≤ 1.5 x upper limit of normal 6. SGOT and SGPT < 2.5 x upper limit of normal 7. Creatinine within institutional normal limits or glomerular filtration rate ≥ 30 mL/min/1.73 m2 by CKD EPI equation (see http://mdrd.com/ for calculator)

9. ECHO: Baseline left ventricular ejection fraction of ≥ 55%

Exclusion Criteria:

1. Pregnant or lactating women. Women of childbearing potential not using a reliable and appropriate contraceptive method. Postmenopausal women must have been amenorrheic for at least 12 months to be considered of non-childbearing potential. Patients of childbearing potential will agree to continue the use of acceptable form of contraception for 24 months from the date of last Herceptin administration.
2. Patients with distant metastasis (brain and/or visceral metastasis)
3. Serious, uncontrolled, concurrent infection(s).
4. Treatment for other carcinomas within the last 5 years, except non-melanoma skin cancer and treated cervical carcinoma in-situ (CCIS)
5. Participation in any investigational drug study within 4 weeks preceding the start of study treatment
6. Other serious uncontrolled medical conditions that the investigator feels might compromise study participation including but not limited to chronic or active infection, HIV-positive patient, uncontrolled hypertension, symptomatic congestive heart failure, unstable angina pectoris, uncontrolled Diabetes mellitus, or psychiatric illness/social situations that would limit compliance with study requirements.
7. Patients with HER2-negative disease

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 53 (Actual)
Dates: Start 2019-11-25 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2026-09-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Olufunmilayo I Olopade, MD, Principal Investigator — University of Chicago
Locations (1):
- University College Hospital, Ibadan, Nigeria, Ibadan, Nigeria

REFERENCES:
- [Derived] Ntekim AI, Ibraheem A, Sofoluwe AA, Kotila O, Babalola C, Karrison T, Olopade CO. ARETTA: Assessing Response to Neoadjuvant Taxotere and Subcutaneous Trastuzumab in Nigerian Women With HER2-Positive Breast Cancer: A Study Protocol. JCO Glob Oncol. 2020 Jul;6:983-990. doi: 10.1200/GO.20.00043. PMID 32628583

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Taxotere and Trastuzumab: Docetaxel/taxotere through drip every 3 weeks for four doses for 12 weeks before a repeat breast ultrasound. After breast ultrasound, if the investigator feels the injection is good, surgery will be done.
  Herceptin/trastuzumab will be given to patients under the skin of the thigh every 3 weeks for 18 times if they are HER2-positive
  Patients with a poor response to docetaxal/herceptin will receive Fluorouracil, Epirubicin Hydrochloride, Cyclophonsphamide (FEC) injection by drip every 3 weeks.
  Hormone-receptor positive patients will receive hormonal therapy with tamoxifen or letrozole after surgery, radiotherapy and LHRH agonist according to the expression of hormone receptors and according to the state of primary menopause at the onset of the study.
  Docetaxel: Administered to all patients for a minimum of 4 cycles for 12 weeks.
  Herceptin: Administered for 18 cycles every three weeks (52 weeks) for each patient starting at the first day of treatment with docetaxel.
  FEC: Only administered to patients who received docetaxel and herceptin and were assessed as having poor response (defined as stable disease or progressive disease or partial response inoperable).
  Tamoxifen: Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  Letrozole: Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  LHRH agonist: Administered to all premenopausal patients.
Period: Overall Study
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Started | 53
Completed | 47
Not Completed | 6
Not completed — Withdrawal by Subject | 4
Not completed — Declined surgery | 2

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
Age, Continuous [Mean (Full Range); unit: years] | 47.6 [25 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  African/Yoruba | 32
  African/Ibo | 9
  African/Other | 6
Region of Enrollment [Number; unit: participants]
  Nigeria | 47

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Complete Pathologic Response (pCR)
Description: Pathological complete response in the breast is defined as the absence of invasive cells at microscopic examination of the primary tumor and lymph nodes at surgery. Any remaining in-situ lesions are permissible. Participants with invalid/missing pCR assessments will be defined as non-responders.
Time Frame: 4-6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
Participants | 25
Statistical Analysis 1: Comparison: Neoadjuvant Taxotere and Trastuzumab; Test type: Superiority; p < 0.001, Exact binomial; Percentage = 53.2, 95% CI 2-sided [38.1 to 67.9]

2. Secondary Outcome: Number of Participants With Adverse Events
Description: Incidence and severity of adverse drug reactions (AE) and serious adverse drug reactions (SAE) including clinical laboratory values, vital signs, ECGs and dose interruptions.
Time Frame: 4-6 months
Measure: Count of Participants; unit: Participants
Groups:
- Neoadjuvant Taxotere and Trastuzumab: Investigators will give patients docetaxel/taxotere through drip every 3 weeks for four doses for 12 weeks before a repeat breast ultrasound. Herceptin/trastuzumab will be given to patients under the skin of the thigh every 3 weeks for 18 times if they are HER2-positive
  Patients with a poor response to docetaxal/herceptin will receive Fluorouracil, Epirubicin Hydrochloride, Cyclophonsphamide (FEC) injection by drip every 3 weeks.
  Hormone-receptor positive patients will receive hormonal therapy with tamoxifen or letrozole after surgery, radiotherapy and LHRH agonist according to the expression of hormone receptors and according to the state of primary menopause at the onset of the study.
  Docetaxel: Administered to all patients for a minimum of 4 cycles for 12 weeks.
  Herceptin: Administered for 18 cycles every three weeks (52 weeks) for each patient starting at the first day of treatment with docetaxel.
  FEC: Only administered to patients who received docetaxel and herceptin and were assessed as having poor response (defined as stable disease or progressive disease or partial response inoperable).
  Tamoxifen: Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  Letrozole: Only administered to hormone-receptor positive patients. Patients will receive tamoxifen or letrozole.
  LHRH agonist: Administered to all premenopausal patients.
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
Participants | 47

3. Secondary Outcome: Progression-free Survival (PFS)
Description: Time from enrollment to disease recurrence or death from any cause.
Time Frame: From start date of therapy to the date of first documented disease progression or death from any cause, whichever may come first, assessed up to 10 years
Reporting Status: Not Posted, anticipated posting 2026-09

4. Secondary Outcome: Duration of Response (DOR)
Description: Time from pathological complete response to disease recurrence or death
Time Frame: Up to 10 years
Reporting Status: Not Posted, anticipated posting 2026-09

5. Secondary Outcome: Analysis of Changes From Baseline Using the Quality of Life (QoL) Instrument: EORTC. Overall Health From Baseline to End of Neoadjuvant Therapy.
Description: Global health status from EORTC QLQ-C30 instrument. Overall health rating on a scale from 1 (very poor) to 7 (excellent). Higher scores indicate better outcome. Values represent changes from baseline with positive values indicating improvement and negative values indicating worsening.
Time Frame: From start date of therapy to end of neoadjuvant therapy approximately 4 - 6 months from commencement of chemotherapy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
units on a scale | -0.57 (0.17)
Statistical Analysis 1: Comparison: Neoadjuvant Taxotere and Trastuzumab; Test type: Other; p = 0.0014, t-test, 2 sided; Paired t-test; Mean Difference (Net) = -0.57, 95% CI 2-sided [-0.91 to -0.24]

6. Secondary Outcome: Analysis of Changes From Baseline Using the Quality of Life (QoL) Instrument: EORTC. Overall Quality of Life From Baseline to End of Neoadjuvant Therapy.
Description: Global quality of life status from EORTC QLQ-C30 instrument. Overall quality of life rating on a scale from 1 (very poor) to 7 (excellent). Higher scores indicate better outcome. Values represent changes from baseline with positive values indicating improvement and negative values indicating worsening.
Time Frame: From start date of therapy to end of neoadjuvant therapy approximately 4 - 6 months from commencement of chemotherapy
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
units on a scale | -0.49 (0.21)
Statistical Analysis 1: Comparison: Neoadjuvant Taxotere and Trastuzumab; Test type: Other; p = 0.023, t-test, 2 sided; Paired t-test; Mean Difference (Net) = -0.49, 95% CI 2-sided [-0.91 to -0.07]

7. Secondary Outcome: Analysis of Changes From Baseline Using the Quality of Life (QoL) Instrument: EORTC. Overall Health From Baseline to 6 Months Post-therapy.
Description: as for outcome 5
Time Frame: From start date of therapy to 6 months post-therapy
Population: Patient completing 6 months of follow-up.
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 37
units on a scale | 0.14 (0.17)
Statistical Analysis 1: Comparison: Neoadjuvant Taxotere and Trastuzumab; Test type: Other; p = 0.44, t-test, 2 sided; Paired t-test; Mean Difference (Net) = 0.14, 95% CI 2-sided [-0.22 to 0.49]

8. Secondary Outcome: Analysis of Changes From Baseline Using the Quality of Life (QoL) Instrument: EORTC. Overall Quality of Life From Baseline to 6 Months Post-therapy.
Description: as for outcome 6
Time Frame: From start date of therapy to 6 months post-therapy
Population: Patient completing 6 months of follow-up
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 37
units on a scale | 0.22 (0.29)
Statistical Analysis 1: Comparison: Neoadjuvant Taxotere and Trastuzumab; Test type: Other; p = 0.46, t-test, 2 sided; Paired t-test; Mean Difference (Net) = 0.22, 95% CI 2-sided [-0.37 to 0.80]

9. Secondary Outcome: Analysis of Changes From Baseline Using the Quality of Life (QoL) Instrument: EORTC
Description: The various domains of QoL over time and the changes from baseline using the validated (by the European Organization for Research and Treatment of Cancer (EORTC)) QoL instrument (global and breast module).
Time Frame: as for outcome 3
Reporting Status: Not Posted, anticipated posting 2026-09

10. Secondary Outcome: Blood Concentrations of Herceptin SC Given in Combination With Docetaxel
Description: Blood concentrations of Herceptin SC at multiple time points using the peak exposure
Time Frame: 21 days
Reporting Status: Not Posted, anticipated posting 2025-12

11. Secondary Outcome: Drug Plasma Concentration of Herceptin SC Given in Combination With FEC
Description: Determine the pharmacokinetic profile of Herceptin SC given in combination with FEC following poor response to TH
Time Frame: 21 days
Reporting Status: Not Posted, anticipated posting 2025-12

12. Secondary Outcome: The Cardiac Toxicity Associated With TscH With FEC +scH in Breast Cancer Patients
Description: The percentage of participants with Heart failure (NYHA Class III or IV or as confirmed by a cardiologist) or a decrease in LVEF of at least 10 EF points from baseline and to below 50%.
Time Frame: Through study completion an average of two years
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
Participants | 1

13. Secondary Outcome: The Cardiac Toxicity Associated With TscH Without FEC +scH in Breast Cancer Patients
Description: The percentage of participants with Heart failure (NYHA Class III or IV or as confirmed by a cardiologist) and a decrease in LVEF of at least 10 EF points from baseline and to below 50%.
Time Frame: Through study completion an average of two years
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
Number analyzed (Participants) | 47
Participants | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | Neoadjuvant Taxotere and Trastuzumab
All-Cause Mortality (participants affected / at risk) | 0/47
Serious Adverse Events (participants affected / at risk) | 7/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Taxotere and Trastuzumab (N=47)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 1
Laboratory abnormality (Investigations) | 1
Hepatobiliary disorders - Other, specify (Hepatobiliary disorders) | 1
Hepatitis viral (Infections and infestations) | 1
Pericardial effusion (Cardiac disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Neoadjuvant Taxotere and Trastuzumab (N=47)
Abdominal pain (Gastrointestinal disorders) | 3
Alanine aminotransferase increased (Investigations) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 34
Anemia (Blood and lymphatic system disorders) | 14
Anorexia (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11
Blood bilirubin increased (Investigations) | 4
Bone pain (Musculoskeletal and connective tissue disorders) | 4
Breast pain (Reproductive system and breast disorders) | 11
Chest pain - cardiac (Cardiac disorders) | 3
Chills (General disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Diarrhea (Gastrointestinal disorders) | 35
Dizziness (Nervous system disorders) | 6
Dry mouth (Gastrointestinal disorders) | 6
Dysphagia (Gastrointestinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3
Edema limbs (General disorders) | 3
Ejection fraction decreased (Investigations) | 3
Fatigue (General disorders) | 6
Febrile neutropenia (Blood and lymphatic system disorders) | 3
Fever (General disorders) | 5
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 17
Headache (Nervous system disorders) | 17
Hot flashes (Vascular disorders) | 5
Hypertension (Vascular disorders) | 3
Hypokalemia (Metabolism and nutrition disorders) | 8
Infusion site extravasation (General disorders) | 3
Injection site reaction (General disorders) | 4
Insomnia (Psychiatric disorders) | 12
Malaise (General disorders) | 8
Mucositis oral (Gastrointestinal disorders) | 3
Nail discoloration (Skin and subcutaneous tissue disorders) | 10
Nausea (Gastrointestinal disorders) | 15
Neutrophil count decreased (Investigations) | 13
Blood and lymphatic system disorders - Other, specify (Blood and lymphatic system disorders) | 8
Cardiac disorders - Other, specify (Cardiac disorders) | 4
Eye disorders - Other, specify (Eye disorders) | 9
Gastrointestinal disorders - Other, specify (Gastrointestinal disorders) | 18
General disorders and administration site conditions - Other, specify (General disorders) | 16
Infections and infestations - Other, specify (Infections and infestations) | 10
Investigations - Other, specify (Investigations) | 12
Metabolism and nutrition disorders - Other, specify (Metabolism and nutrition disorders) | 4
Musculoskeletal and connective tissue disorder - Other, specify (Musculoskeletal and connective tissue disorders) | 28
Nervous system disorders - Other, specify (Nervous system disorders) | 7
Reproductive system and breast disorders - Other, specify (Reproductive system and breast disorders) | 5
Respiratory, thoracic and mediastinal disorders - Other, specify (Respiratory, thoracic and mediastinal disorders) | 4
Skin and subcutaneous tissue disorders - Other, specify (Skin and subcutaneous tissue disorders) | 25
Pain (General disorders) | 10
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5
Palpitations (Cardiac disorders) | 3
Paresthesia (Nervous system disorders) | 3
Peripheral motor neuropathy (Nervous system disorders) | 5
Peripheral sensory neuropathy (Nervous system disorders) | 12
Platelet count decreased (Investigations) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 6
Rash acneiform (Skin and subcutaneous tissue disorders) | 6
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 4
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 17
Skin ulceration (Skin and subcutaneous tissue disorders) | 3
Sore throat (Respiratory, thoracic and mediastinal disorders) | 5
Stomach pain (Gastrointestinal disorders) | 3
Upper respiratory infection (Infections and infestations) | 4
Vaginal infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 17
Watering eyes (Eye disorders) | 6
White blood cell decreased (Investigations) | 14

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-30): https://cdn.clinicaltrials.gov/large-docs/77/NCT03879577/Prot_SAP_000.pdf